CLINICAL TRIAL: NCT04904900
Title: Prospective Evaluation of a Fast-track Treatment Pathway for Patients With Chronic Hepatitis B Under Primary Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lai Hung Wong, Professor, Chinese University of Hong Kong
Other Study IDs: HBV_GOPC study
Record Dates: First submitted 2021-05-20; First posted 2021-05-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Chronic Hep B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample for
  * Liver function test (including albumin, bilirubin, ALT)
  * Alpha-fetoprotein
  * Hepatitis B surface antigen (HBsAg), Hepatitis B e antigen (HBeAg) and antibody to Hepatitis B e antigen (anti-HBe)
  * HBV DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective-prospective longitudinal cohort study, with analyses performed before and after introduction of the pathway, and comparisons made to unexposed controls. We will launch a protocol-driven management for CHB patients, and provide the appropriate assessment tools (transient elastography, HBV DNA assay) to general outpatient clinics (GOPC) in Hong Kong. Patients who fulfil treatment criteria will be referred to specialist outpatient clinics (SOPC) in a fast-track manner. We will also evaluate the linkage-to-care rate 3 years before the launch of this care pathway retrospectively.

DETAILED DESCRIPTION:
Chronic viral hepatitis is the seventh leading cause of mortality globally, responsible for 1.45 million deaths in 2013. The consequences of chronic hepatitis B and C infection - cirrhosis and liver cancer - account for 94% of deaths associated with hepatitis.1 Liver cancer is the second most common cause of cancer death in the Asia-Pacific region. Approximately 78% of liver cancer cases are a result of chronic viral hepatitis.1,2 In Hong Kong, the positive rate of hepatitis B surface antigen (HBsAg) remains high among adults of productive ages of 31-40 and 41-50 years (5.2% and 7.2% respectively) in 2015.3 World Health Organization (WHO) published the first global health sector strategy on viral hepatitis in June 2016, a strategy that contributes to the proposed targets for the reduction of chronic viral hepatitis incidence and mortality of 90% and 65% respectively by 2030.4 The Chief Executive's 2017 Policy Address in Hong Kong asked to set up the Steering Committee to formulate strategies to effectively prevent and control viral hepatitis.5 The Steering Committee is currently reviewing local and international trends and developments in the prevention and control of viral hepatitis; advising the Government on policies and cost-effective targeted strategies for prevention and control of viral hepatitis; and conducting and coordinating the surveillance and evaluation of viral hepatitis control and recommending appropriate response.5 One of the key gaps in CHB management is the suboptimal treatment in patients who fulfil treatment criteria but not started on antiviral treatment because of linkage-to-care issue, namely very long waiting time (up to 2.5 years) from primary care setting like general outpatient clinics (GOPC). There are limited resources for specialized assessments (e.g. HBV DNA assays, transient elastography for liver fibrosis assessment).

Therefore a novel fast-track treatment pathway for patients with chronic hepatitis B under primary care would fill this gap and provide pivotal data to the Government and the Steering Committee to guide the strategies for achieving the goals set by WHO.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with positive hepatitis B surface antigen (HBsAg) for 6 months
* Under the care of GOPC

Exclusion Criteria:

* Age under 18
* Refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 prospectively from FM/GOPC 3000 retrospectively from CDARS.
Sampling Method: Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Linkage-to-care | 3 years
  referral rate of patients from GOPC and SOPC who fulfil treatment criteria

SECONDARY OUTCOMES:
Unnecessary referral | 3 years
  referral rate of patients from GOPC and SOPC who do not fulfil treatment criteria
GOPC care management rate | 3 years
  transient elastography uptake rate, fibrosis staging, clinical events, default rate
SOPC care management rate | 3 years
  antiviral uptake care, fibrosis staging, clinical events, default rate

CONTACTS AND LOCATIONS:
Overall Officials: Grace LH Wong, Prof, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- See also: Hepatitis B — http://www.who.int/en/news-room/fact-sheets/detail/hepatitis-b
- See also: Hepatitis C — http://www.who.int/en/news-room/fact-sheets/detail/hepatitis-c
- See also: Surveillance of Viral Hepatitis in Hong Kong - 2016 Update Report — https://www.chp.gov.hk/files/pdf/viral_hepatitis_report_2016_final.pdf
- See also: Combating hepatitis B and C to reach elimination by 2030 — https://www.who.int/publications/i/item/combating-hepatitis-b-and-c-to-reach-elimination-by-2030
- See also: Building a Caring, Inclusive Society, Improving People's Livelihood — https://www.policyaddress.gov.hk/2017/eng/pdf/Agenda_Ch6.pdf